CLINICAL TRIAL: NCT00238836
Title: Anticipatory & Preventive Team Care (APTCare): At Risk Patients of Family Health Networks
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: C. T. Lamont Primary Care Research Centre (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); University of Ottawa (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APTCare
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2005-06

CONDITIONS: Diabetes; Chronic Obstructive Pulmonary Disease; Congestive Heart Failure; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive; Heart Failure; Hypertension

INTERVENTIONS:
Behavioral: Self-management of chronic illness

SUMMARY:
The University of Ottawa and Élisabeth Bruyère Research Institute are conducting a study of preventive care for frail patients at risk of functional decline. At risk patients are assigned by chance to continue receiving their standard care from their family physician or receive additional care from a nurse practitioners and a pharmacist. In collaboration with the family physician, they develop an individualized care plan, a treatment and management road plan, for each patient, which they implement over the study period of one approximately year. The objective of the study is to compare the effectiveness of the model of care that includes the nurse practitioners and pharmacist against standard care in preventing functional decline, to determine the acceptability of this model of care to patients, their caregivers and the medical team, and to evaluate the cost implication of the program.

ELIGIBILITY:
Inclusion Criteria:

* 50 years and over
* 'At Risk' by having one or more of the following: a. Visits to emergency dept within the past 6 months; b. Admission to hospital for a medical problem in past 6 months; c. High service use profiles; d. Polypharmacy; e. Other high risk factors
* Capable of giving informed consent
* Able to use the Care Companion technology

Exclusion Criteria:

* Cognitive impairment such that they cannot give informed consent
* Unable or unwilling to use the telehomecare equipment
* Unlikely to tolerate the intensive intervention
* Language or cultural barriers
* Being acutely ill or having an unstable condition on entry to the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: William Hogg, MD, Principal Investigator — C. T. Lamont Primary Care Research Centre; Jacques Lemelin, MD, Principal Investigator — University of Ottawa
Locations (1):
- West Carleton Family Health Network, Carp, Ontario, Canada

REFERENCES:
- [Derived] Fletcher J, Hogg W, Farrell B, Woodend K, Dahrouge S, Lemelin J, Dalziel W. Effect of nurse practitioner and pharmacist counseling on inappropriate medication use in family practice. Can Fam Physician. 2012 Aug;58(8):862-8. PMID 22893340
- [Derived] Dahrouge S, Hogg W, Lemelin J, Liddy C, Legault F. Methods for a study of Anticipatory and Preventive multidisciplinary Team Care in a family practice. Can Fam Physician. 2010 Feb;56(2):e73-83. PMID 20154234
- [Derived] Gray D, Armstrong CD, Dahrouge S, Hogg W, Zhang W. Cost-effectiveness of Anticipatory and Preventive multidisciplinary Team Care for complex patients: evidence from a randomized controlled trial. Can Fam Physician. 2010 Jan;56(1):e20-9. PMID 20090057
- [Derived] Hogg W, Lemelin J, Dahrouge S, Liddy C, Armstrong CD, Legault F, Dalziel B, Zhang W. Randomized controlled trial of anticipatory and preventive multidisciplinary team care: for complex patients in a community-based primary care setting. Can Fam Physician. 2009 Dec;55(12):e76-85. PMID 20008582